CLINICAL TRIAL: NCT00268281
Title: Left Ventricular Capture Management (LVCM) Software Download Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 238
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Heart Failure
Keywords: cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Left Ventricular Capture Management Software

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy (CRT) may be prescribed.

Left Ventricular Capture Management (LVCM) refers to the overall method for determining left ventricular thresholds (level of energy needed to effectively pace the tissue in the lower left chamber of the heart) by measuring, analyzing, and adjusting energy delivered from the CRT device to the pacing lead.

The purpose of the Left Ventricular Capture Management Software Download Clinical Trial was to evaluate the accuracy of the Left Ventricular Capture Management (LVCM) feature to support LVCM feature approval in future cardiac resynchronization therapy with defibrillation (CRT-D) devices

ELIGIBILITY:
Inclusion Criteria:

* Subjects who successfully underwent implantation of an InSync II Marquis system

Exclusion Criteria:

* Subjects who are post-heart transplant
* Subjects enrolled in a concurrent study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107
Dates: Start 2004-12; Study Completion 2005-07

PRIMARY OUTCOMES:
To evaluate the accuracy of left ventricular capture management (LVCM)

SECONDARY OUTCOMES:
To compare left ventricular capture management (LVCM) measurements to a similar measurement taken automatically when subjects are completing normal daily activities
To evaluate subject rhythm and rate immediately following an LVCM measurements
To characterize all adverse events

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Palo Alto, California
  - Bridgeport, Connecticut
  - Atlantis, Florida
  - Ormond Beach, Florida
  - Oak Lawn, Illinois
  - Indianapolis, Indiana
  - Portland, Maine
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - West Orange, New Jersey
  - Charlotte, North Carolina
  - Wynnewood, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Richmond, Virginia
  - Morgantown, West Virginia